CLINICAL TRIAL: NCT00049114
Title: A Phase I-II Study of R115777 (ZARNESTRA) Plus Doxorubicin and Cyclophosphamide in Patients With Locally Advanced Breast Cancer and Metastatic Breast Cancer
Brief Title: Tipifarnib, Doxorubicin, and Cyclophosphamide in Treating Women With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02500; 02-05-125; AECM-0205125; NCI-5598; CDR0000257811; N01CM62204 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Inflammatory Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; tipifarnib; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (doxorubicin, cyclophosphamide, tipifarnib, G-CSF) (Experimental): PHASE I (nonregional stage IV disease) (closed to accrual as of 1/19/04): Patients receive doxorubicin IV over 10-15 minutes and cyclophosphamide IV over 30 minutes on day 1, oral tipifarnib twice daily on days 2-7, and G-CSF subcutaneously on days 2-13. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  PHASE II (stage IIB, IIIA, IIIB, or IIIC): Patients receive tipifarnib at the MTD and doxorubicin, cyclophosphamide, and G-CSF as in phase I (phase I closed to accrual as of 1/19/04). After the fourth course, patients may undergo complete resection.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Drug: tipifarnib; Biological: filgrastim; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: doxorubicin hydrochloride
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen
Procedure: therapeutic conventional surgery — Undergo complete resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as doxorubicin and cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining tipifarnib with doxorubicin and cyclophosphamide may kill more tumor cells. Phase II trial to study the effectiveness of combining tipifarnib with doxorubicin and cyclophosphamide in treating women who have locally advanced breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of tipifarnib when administered with doxorubicin and cyclophosphamide in women with metastatic breast cancer (non-regional stage IV disease). (Phase I closed to accrual as of 1/19/04) II. Determine the pathologic complete remission rate in patients with locally advanced breast cancer (stages IIB, IIIA, IIIB, or IIIC) treated with the recommended phase II dose of this regimen.

SECONDARY OBJECTIVES:

I. Determine the clinical complete response rate in patients treated with this regimen.

II. Determine the toxicity profile of this regimen in these patients. III. Correlate pretreatment levels of ErbB1, 2, 3, 4 and phosphorylated levels of Akt, STAT3, and Erk ½ with clinical response in these patients and with percent inhibition of proliferation (Ki-67) and percent induction of apoptosis in post-treatment tumor specimens.

IV. Correlate percent decrease of farnesyltransferase (FTase) activity levels, HDJ-2 farnesylation, phospho-Akt, phospho-STAT3, and phospho-Erk ½ with clinical response rates in these patients and with percent inhibition of proliferation (Ki-67) and percent inhibition of apoptosis.

OUTLINE: This is a multicenter, dose-escalation study of tipifarnib. Patients are stratified according to presence of inflammatory carcinoma (yes vs no).

PHASE I (nonregional stage IV disease) (closed to accrual as of 1/19/04): Patients receive doxorubicin IV over 10-15 minutes and cyclophosphamide IV over 30 minutes on day 1, oral tipifarnib twice daily on days 2-7, and filgrastim (G-CSF) subcutaneously on days 2-13. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II (stage IIB, IIIA, IIIB, or IIIC): Patients receive tipifarnib at the MTD and doxorubicin, cyclophosphamide, and G-CSF as in phase I (phase I closed to accrual as of 1/19/04). After the fourth course, patients may undergo complete resection.

Patients are followed every 3-4 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 3-12 patients will be accrued for phase I (closed to accrual as of 1/19/04) of this study. A total of 21-50 patients will be accrued for phase II of this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast
* Phase I (closed to accrual as of 1/19/04):

  * Nonregional stage IV disease
* Phase II:

  * Locally advanced disease, according to AJCC staging criteria:

    * Stage IIB
    * Stage IIIA
    * Stage IIIB
    * Stage IIIC
* At least 1 bidimensionally or unidimensionally measurable indicator lesion
* Hormone receptor status:

  * Not specified
* Female
* Performance status - ECOG 0-1
* Performance status - Karnofsky 70-100%
* Not specified
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* LVEF normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No other invasive malignancies within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to tipifarnib or other agents used in the study (e.g., imidazoles or quinolones)
* No ongoing or active infection
* No other concurrent uncontrolled illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not specified
* Phase I (closed to accrual as of 1/19/04):

  * More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
  * No more than 1 prior adjuvant/neoadjuvant regimen and 1 prior regimen for metastatic disease
  * Prior doxorubicin allowed provided the following are true:

    * Used in adjuvant setting
    * Cumulative dose was no greater than 240 mg/m^2
    * At least 1 year between completion of adjuvant therapy and relapse
* Phase II:

  * No prior chemotherapy for locally advanced breast cancer
* At least 1 week since prior tamoxifen or other selective estrogen receptor modulators for prevention or other indications (e.g., osteoporosis, ductal carcinoma in situ, or invasive breast cancer)
* Phase I (closed to accrual as of 1/19/04):

  * More than 4 weeks since prior radiotherapy
* Phase II:

  * No prior radiotherapy for locally advanced breast cancer
* Not specified
* No antacids within 2 hours of study drug administration
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-02; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Pathological complete response in the breast | 8 weeks
  95% confidence intervals of these estimates will be obtained.

SECONDARY OUTCOMES:
Proportion of patients who have a clinical complete response | 8 weeks
  95% confidence intervals of these estimates will be obtained.
Grade 3 or 4 toxicities assessed using NCI CTCAE version 3.0 | Up to 5 years
  Toxicity will be summarized by type, frequency and severity. This will be compared with an historical database.
Median disease-free survival | Up to 5 years
  Will be summarized, and 95% confidence intervals of these estimates will be obtained.
Percentage of patients free of disease | 1 year
  Will be summarized, and 95% confidence intervals of these estimates will be obtained.
Percentage of patients free of disease | 2 years
  Will be summarized, and 95% confidence intervals of these estimates will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sparano, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States